CLINICAL TRIAL: NCT05323578
Title: Consumption Status of Caffeine and Adverse Effects Experience Among Anesthetists
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Raham Hasan Mostafa, MD, Assistant Professor of Anesthesia, Ain Shams University
Other Study IDs: R 66/2022
Record Dates: First submitted 2022-04-05; First posted 2022-04-12 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Caffeine; Caffeine Withdrawal; Caffeine Dependence
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — Prevalence of safe caffeine consumption among anesthetists

SUMMARY:
High-caffeine consumption has been increasing in physicians, frequently causing the most common symptoms such as tremor, insomnia, anxiety, and nervousness and rarely leading to serious adverse effects like seizure, acute mania, and stroke due to caffeine overdose. There have been no studies regarding analysis of high-caffeine consumption and its adverse effects among anesthetists.

DETAILED DESCRIPTION:
This study was to examine high-caffeine consumption patterns, associated factors, and adverse effects based on responses anesthetists with different age of experience.

ELIGIBILITY:
Inclusion Criteria:

* Any anesthetist

Exclusion Criteria:

* Pregnancy

Ages: 24 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Almost all anesthetists who approved to continue the survey.
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
The prevalence of caffeine consumption among a sample of anesthesiologists, to determine their caffeine daily intake in relation to the safe level suggested by the European Food Safety Authority (EFSA). | 24 hours
  Average daily amount of caffeine consumption in mg
Subgroup comparison between junior and senior anesthetists | 24 hours
  Average daily amount of caffeine consumption in mg

CONTACTS AND LOCATIONS:
Overall Officials: Raham H Mostafa, MD, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
The datasets used and/or analyzed during the current study are available from the corresponding author on reasonable request